CLINICAL TRIAL: NCT00488670
Title: An Open-label Study of Escitalopram in the Treatment of Major Depressive Disorder in Elderly Patients With Alzheimer's Disease
Brief Title: Escitalopram and Depression in Elderly Alzheimer's Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Dr. Rabheru left VCH last year and the study was cancelled according to his research coordinator.
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Kiran Rabheru, University of British Columbia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H07-00050
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-06

CONDITIONS: Depressive Disorder
Keywords: Alzheimer's disease; elderly; open-label; escitalopram
MeSH Terms: conditions — Depressive Disorder; Alzheimer Disease | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Escitalopram — See Detailed Description.

SUMMARY:
To investigate the effect of Escitalopram in a large and diverse of dementia patients suffering from depression.

DETAILED DESCRIPTION:
This study will assess the efficacy, tolerability, and safety of escitalopram in the treatment of Major Depressive Disorder in patients with Alzheimer's disease over a 24-week period. It will also assess the efficacy and tolerability of escitalopram after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* > 50 years
* Male & female
* Alzheimer's disease
* Depressive episode

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in Cornell Scale for Depression in Dementia (CSDD) from baseline.

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale; Neuropsychiatric Inventory; Alzheimer's Disease Cooperative Study

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Rabheru, MD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Mt. St. Joseph's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia